CLINICAL TRIAL: NCT03419416
Title: KMC Implementation Research for Accelerating Scale-up in Oromia Region, Ethiopia
Acronym: KMC-Oromia
Status: Completed | Type: Observational
Sponsor: Addis Ababa University (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Damen Haile Mariam, Prof. Damen Haile Mariam, Addis Ababa University
Other Study IDs: 201523748
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Low Birth-weight
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kangaroo mother care (KMC) — Skin to skin contact of newborns with mothers and exclusive breast feeding

SUMMARY:
The main objective is to implement Kangaroo Mother Care (KMC) at selected facilities in Addis Ababa and Oromia Regions to achieve high effective coverage in the catchment population.

DETAILED DESCRIPTION:
To achieve the objective summarized above, the investigators will engage in an iterative process using program learning and quantitative data to continuously improve models in order to enhance uptake of KMC in two phases.

In phase 1, the model will undergo an iterative process whereby every three months, the investigators will analyze the data collected and improve the model until it is reached at a model that achieves effective KMC coverage of at least 80%.

In phase 2, we will scale the successful model to all selected facilities.

The investigators' primary outcomes will be effective coverage of KMC at 7 days of age, and effective coverage of KMC at 7 days after discharge from the facility. Effective coverage will be defined as adoption of skin to skin care for at 8 least hours and exclusive breastfeeding in the 24 hours prior to assessment

ELIGIBILITY:
Inclusion Criteria:

* All newborns who are less than 2000 gm born within the study facilities during the study period.

Exclusion Criteria:

* Newborns who are sick per predefined criteria will not be provided KMC until they have been stabilized. Criteria for delay of initiation include: critical illness including apnea, decreased respiratory rate <20 breaths per minute, grunting, cyanosis, severe chest in-drawing, convulsions, unconsciousness, and severe hypothermia <32°F.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be low birth weight babies (less than 2000 gm) within the study sites. The study sites are one primary hospital in Addis Ababa Region and two primary and one referral hospital in Oromia Region.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Effective coverage of KMC at 7 days of age. | Seven days of age
  Effective coverage will be defined as adoption of skin-to-skin care for at least 8 hours and exclusive breastfeeding in the 24 hours prior to assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Bahl, MD, PhD, Study Director — World Health Organization
Locations (2):
- Ethiopia (2):
  - Tirunesh Beijing Hospital, Akaki, Addis Ababa
  - Batu Hospital, Ādamī Tulu, Oromiya

REFERENCES:
- [Derived] Mony PK, Tadele H, Gobezayehu AG, Chan GJ, Kumar A, Mazumder S, Beyene SA, Jayanna K, Kassa DH, Mohammed HA, Estifanos AS, Kumar P, Jadaun AS, Hailu Abay T, Washington M, W/Gebriel F, Alamineh L, Fikre A, Kumar A, Trikha S, Ashebir Gebregizabher F, Kar A, Bilal SM, Belew ML, Debere MK, Krishna R, Dalpath SK, Amare SY, Mohan HL, Brune T, Sibley LM, Tariku A, Sahu A, Kumar T, Hadush MY, Gowda PD, Aziz K, Duguma D, Singh PK, Darmstadt GL, Agarwal R, Gebremariam DS, Martines J, Portela A, Jaiswal HV, Bahl R, Rao Pn S, Tadesse BT, Cranmer JN, Hailemariam D, Kumar V, Bhandari N, Medhanyie AA; KMC Scale-Up Study Group. Scaling up Kangaroo Mother Care in Ethiopia and India: a multi-site implementation research study. BMJ Glob Health. 2021 Sep;6(9):e005905. doi: 10.1136/bmjgh-2021-005905. PMID 34518203
- [Derived] Medhanyie AA, Alemu H, Asefa A, Beyene SA, Gebregizabher FA, Aziz K, Bhandari N, Beyene H, Brune T, Chan G, Cranmer JN, Darmstadt G, Duguma D, Fikre A, Andualem BG, Gobezayehu AG, Mariam DH, Abay TH, Mohan HL, Jadaun A, Jayanna K, Kajal FNU, Kar A, Krishna R, Kumar A, Kumar V, Madhur TK, Belew ML, M R, Martines J, Mazumder S, Amin H, Mony PK, Muleta M, Pileggi-Castro C, Pn Rao S, Estifanos AS, Sibley LM, Singhal N, Tadele H, Tariku A, Lemango ET, Tadesse BT, Upadhyay R, Worku B, Hadush MY, Bahl R; KMC Scale-Up Study Group. Kangaroo Mother Care implementation research to develop models for accelerating scale-up in India and Ethiopia: study protocol for an adequacy evaluation. BMJ Open. 2019 Nov 21;9(11):e025879. doi: 10.1136/bmjopen-2018-025879. PMID 31753865